CLINICAL TRIAL: NCT06455384
Title: The Genetics Navigator: Evaluating a Digital Platform for Genomics Health Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4033
Record Dates: First submitted 2023-09-05; First posted 2024-06-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Conditions; Connective Tissue Diseases; Retinal Disease; Epilepsy in Children; Neurodevelopmental Disorders; Cancer; Polyposis
Keywords: Genomic Sequencing; Randomized Controlled Trial; Clinical Utility; Personal Utility; Decision Aid; Incidental Findings
MeSH Terms: conditions — Connective Tissue Diseases; Retinal Diseases; Neurodevelopmental Disorders; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetics Navigator (Experimental): Participants in the intervention arm will use the Genetics Navigator to support the delivery of genetic services, including intake, education, pre- and post-test counselling, return of results, and physician-generated management recommendations. Participants in the experimental arm will also receive standard of care genetics care.
  Interventions: Behavioral: Genetics Navigator
- Standard Care with Genetics Professionals (Active Comparator): Participants in the control arm will receive their genetic counselling and test results through usual care, which consists of in-person/phone/video-conference consults with genetic counsellors and medical geneticists.
  Interventions: Behavioral: Standard Care with Genetics Professionals

INTERVENTIONS:
Behavioral: Genetics Navigator — The Genetics Navigator will be used to support patients during the delivery of genetic services, including intake, education, pre- and post-test counselling, and physician-generated management recommendations
  Arms: Genetics Navigator
Behavioral: Standard Care with Genetics Professionals — Standard care for the delivery of genetic services, including receiving genetic counselling and test results
  Arms: Standard Care with Genetics Professionals

SUMMARY:
Genetic testing (GT) (including targeted panels, exome and genome sequencing) is increasingly being used for patient care as it improves diagnosis and health outcomes. In spite of these benefits, genetic testing is a complex and costly health service. This results in unequal access, increased wait times and inconsistencies in care. The use of e-health tools to support genetic testing delivery can result in a better patient experience and reduced distress associated with waiting for results and empower patients to receive and act on medical results. We have previously developed and tested an interactive, adaptable and patient-centred digital decision support tool (Genetics ADvISER) to be used for genetic testing decision making, and have now developed the Genetics Navigator (GN), a patient-centred e-health navigation platform for end-to-end genetic service delivery. The objective of this study is to evaluate the effectiveness of the GN in an RCT in reducing distress with patients and parents of patients being offered genetic testing. Results of this trial will be used to establish whether the GN is effective to use in practice. If effective, GN could fill a critical clinical care gap and improve health outcomes and service use by reducing counselling burden as well as overuse, underuse and misuse of services. These are concerns policy makers seek to address through the triple aims of health care1. This study represents a significant advance in personalized health by assessing the effectiveness of this novel, comprehensive e-health platform to ultimately improve genetic service delivery, accessibility, patient experiences, and patient outcomes.

DETAILED DESCRIPTION:
BACKGROUND: Genetic testing is a catalyst for personalized health. Technologies such as targeted panels and genomic sequencing (GS) are exerting a profound influence on clinical care by ushering personalized medicine into mainstream practice. With substantial improvements in diagnostic performance has come unprecedented demand for genetic testing for a broad range of clinical indications.The volume of testing and complexity of genetic testing analysis places unsustainable pressure on the standard model of care for delivering genetics services, which is heavily dependent on multiple interconnected clinical specialists including medical geneticists, genetic counsellors, clinical laboratory directors, bioinformaticians, and genome analysts based in tertiary care centres. With this increased demand, innovative strategies for increasing capacity and efficiency of genetic service delivery are needed. Our research team has built on our previous preliminary work to develop the Genetics Navigator (GN) to fill this gap. The GN is meant to provide end-to-end support to genomic services and patients who are offered genetic testing. The GN is meant to provide patients with information about genetic testing, help patients make decisions about genetic testing, collect patient history and family history collection before their appointment, and provide genetic test results. The study is interested in comparing the effectiveness of the Genetics Navigator with traditional medical appointments with genetic counsellors and medical geneticists.

RATIONALE: There are limited e-health tools for the delivery of GS. Few e-health tools exist to support the comprehensive delivery of GS and very few have been rigorously evaluated.61 Existing tools target cancer settings,42 education36 or return of results46 but are not integrated to enable a seamless end-to-end patient journey. Consequently, existing tools are limited in scope and scale. Finally, due to the lack of comprehensive e-health tools for GS, little is known about end users' needs for an e-health platform. Understanding end users' needs and requirements are critical to the development of an effective e-health solution for GS health service delivery. Finally, the development of our Genetics Navigator tool represents an innovative strategy to address significant health service delivery barriers and advance the implementation of personalized health by increasing efficiency of genetic service delivery and improving patient experience.

OBJECTIVES AND HYPOTHESIS: Evaluate the effectiveness, cost-effectiveness, and user experience of the Genetics Navigator compared to usual care (standard genetic counselling) with patients and parents of patients receiving genetic testing. Hypothesis: Use of the Genetics Navigator will improve emotional functioning (decrease distress [primary outcome], anxiety, and decisional conflict), knowledge, quality of life, patient empowerment, personal utility, and intention to and actual follow through with management recommendations compared to usual care.

METHOD: This is a non-blinded prospective repeated measures randomized controlled superiority trial where we will evaluate the effectiveness and cost-effectiveness of the Genetics Navigator in reducing patient distress compared to usual care. As a part of this trial, patients will receive genetic test results related to a range of clinical indications. A qualitative sub-study will examine user experience.

STUDY POPULATION:

Trial: Adult genetics patients (aged ≥18 years) at Sinai Health System (Sinai) and parents/legal guardians of pediatric patients at the Hospital for Sick Children (SickKids) who are currently eligible to receive clinical genetic testing, as determined by a medical geneticist.

Qualitative Interviews: We will interview a purposive sample of up to 20 adult patients and 20 parents/ legal guardians in each arm within 6 months of completing their participation.

INTERVENTION: Participants in the intervention arm will use the Genetics Navigator to support the delivery of genetic services, including intake, education, pre- and post-test counselling, and physician-generated management recommendations. The Navigator will be supported by consults with genetics professionals via in-person/phone/video-conferencing.

CONTROL:Participants in the control arm will receive their genetic counselling and test results through usual care, which consists of in-person/phone/video-conference consults with genetic counsellors and medical geneticists.

ELIGIBILITY:
Inclusion:

* Adult patients (18 years of age or older) who are referred to participating clinicians at Mount Sinai Hospital for clinical genetic testing.
* Parents/legal guardians (18 years of age or older) of pediatric patients who are referred to participating clinicians at SickKids for clinical genetic testing.

Exclusion:

* Known not to be eligible for clinical genetic testing in Ontario
* Requires urgent clinical genetic testing or prenatal genetic testing
* Not fluent in English (speaking and reading)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Multi-Dimensional Impact of Cancer Risk Assessment (MICRA) | At 6 months and 9 months after baseline
  The Multi-Dimensional Impact of Cancer Risk Assessment (MICRA) is a 25-item standardized, validated scale that measures the impact of result disclosure from genetic tests. There are three subscales: Distress (6 items), Uncertainty (9 items) and Positive Experiences (4 items). Total scores range from 0-125, with higher scores indicating worse outcome. Scores on the Distress subscale range from 0-30, with higher scores indicating worse outcome. Scores on the Uncertainty subscale range from 0-45, with higher scores indicating worse outcome. Scores on the Positive Experiences Subscale range from 0-20, with higher scores indicating worse outcomes. (PMID: 12433008)

SECONDARY OUTCOMES:
University of North Carolina Genomic Knowledge Scale (UNC-GKS) | Assessed at baseline, 2 weeks, 1 month, 6 months and 9 months
  Knowledge is measured using the Genomic Knowledge Scale developed by The University of North Carolina. The scale is an established scale measuring genomics knowledge. Patients mark 25 statements about genes, genetic effects on health, familial inheritance, and diagnostic exome sequencing. Respondents mark each as true, false, or not sure/don't know (scored as incorrect). Correct responses are scored as 1 and summed. Possible scores range from 0-25. Higher scores indicates a higher level of knowledge (PMID: 29928697).
SURE | Assessed at 1 month
  The SURE screening test is a 4-item tool to assess decisional conflict in patients, developed by Légaré et al. Each item is scored as a yes (1) or no (0), and a total score is calculated by summing all items. A score less than 4 indicates the probability that a patient experiences clinically significant decisional conflict.
Hospital Anxiety and Depression Scale (HADS) | Assessed at baseline, 2 weeks, 1 month, 6 months and 9 months
  Measured using the 14 item scale, each item is answered on a four point (0-3) response category. Possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression. Items can be summed and scored for both depression and anxiety, with a score above 11 indicates a case (depression or anxiety).
The Genomics Outcome Scale (GOS) | Assessed at 2 weeks, 1 month, 6 months and 9 months
  Patient empowerment is measured using the a shorter version of the Genetic Counselling Outcome Scale (GCOS-24), called Genomics Outcome Scale (GOS). The scale uses 6 patient reported outcome measure items to evaluate genetic counselling and testing services. Each item is scored on a 5-point scale and the final score is calculated by summing all items. Each of the 6 items in the measure is rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree) with possible total scores ranging from 6 to 42. A higher score indicates greater empowerment. (PMID: 30496830)
36-item Short Form Survey (SF-36) | Assessed at baseline, 2 weeks, 1 month, 6 months and 9 months
  The SF-36 scale measures quality of life. The SF-36 has 36 items that address physical and mental functioning. Physical and mental health composite scores range from 0 to 100, with 0 indicating the lowest possible level of health, and 100 indicating the highest possible level of health.
Satisfaction with Decision Making Scale | Assessed at 1 month
  A six item scale measures a patient satisfaction with a health care decision. Items are scored 1-4. A higher score signifies a higher level of satisfaction or preparation with a decision. Items can be summed and scored (sum the 6 items and divide by 6).
Preparation for Decision Making Scale | Assessed at 1 month
  A 10 item scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation visit and making a health decision. Items are scored 1-4. Items can be summed and scored (sum the 10 items and divide by 10). A higher score indicates a higher level of preparation.
Acceptability e-Scale | Assessed at 2 weeks, 1 month, 6 months and 9 months
  The 6 item Acceptability E-Scale measures acceptability and usability of the platform. The AES includes dimensions of ease of use, understandability of questions, enjoyability of experience, whether the length of time is acceptable, helpfulness, and overall satisfaction, using a 5-point response scale for each item (1=not acceptable, 5=highly acceptable). Scores range from 6 to 30 with a higher score indicating higher acceptability.
Digital Health Literacy Scale (DHLS) | Control: Assessed at baseline; Intervention: Assessed at baseline
  Digital Health Literacy Scale (DHLS) is a 3 item scale that measures a respondent's perceived skill at using and applying electronic information technology to health problems. Each item is on a five-point Likert scale ranging from strongly agree to strongly disagree, with responses being assigned a value of 0-4. The scores range from 0-12 with higher scores indicating higher digital health care literacy.
Frequency of platform use | Baseline
  Measure of the amount of times the digital platform was accessed by the participant.
Duration of platform session | 2 weeks, 6 months and 9 months
  Measure of total time spent using the digital platform.
Answers to platform questions | Assessed at 2 weeks, 6 months and 9 months
  Measure of value preferences, preference lean and preparation for results.
Duration of genetic counselling session | Control: immediately after pre-test meeting with clinician, immediately after post-test meeting with clinician; Intervention: immediately after pre-test meeting with clinician, immediately after post-test meeting with clinician
  Measure of total time spent with Genetic counselor in the counselling session.
Qualitative outcomes of counselling sessions | 2 weeks and 6 months
  Patients pre- and post-test clinical encounters will be assessed based off of medical chart notes.
Qualitative interviews with a subset of participants and providers | 9 months
  We will use in-depth interviews with patients to provide further insights into the delivery and support of genetic services. Interviews will consider participants' socio-demographic factors that may influence their informational, decisional, and follow-up needs as well as how they engage with genetic information, participate in shared decision making, and manage genetic test results. The qualitative analyses for the interviews will draw on grounded theory. We will use open coding, constant comparison and axial coding to identify common and divergent themes to characterize the entire dataset. Two researchers will code transcripts independently; consensus on codes will be reached through discussion. Validation methods may include triangulation and member checking. In keeping with qualitative methodology, data analysis will occur in conjunction with data collection. On-going analysis will inform the development of progressive iterations of the interview guides.
BRIEF Health Literacy Screening Tool (BRIEF) | Assessed at baseline
  BREIF is a 4-item scale used to assess health literacy. Each item is quantified using a 5-point scale (1-5) with higher scores indicating higher health literacy.
Health Resource Use Questionnaire (RUQ) | Assessed at 1 month and 9 months
  This survey was developed to learn more about the resources related to health, social and community services used to reduce stress of anxiety related to coping with a patient's condition. This is not a scale, each items reports descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Bombard, PhD, Principal Investigator — St. Michael's Hospital and University of Toronto; Robin Hayeems, PhD, Principal Investigator — The Hospital for Sick Children and University of Toronto
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Sunnybrook Hospital, Toronto

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to research who are interested in / conducting similar research in this field. This data will be available upon request, keeping with research ethics procedures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For 5 years after study has been completed and the trail data has been published.
Access Criteria: Data will be made available to research who are interested in / conducting similar research in this field. This data will be available upon request, keeping with research ethics procedures.
URL: https://research.unityhealth.to/labs/yvonne-bombard/

REFERENCES:
- [Derived] D'Amours G, Clausen M, Luca S, Reble E, Kodida R, Assamad D, Bernier F, Chad L, Costain G, Dhalla I, Faghfoury H, Friedman JM, Hewson S, Jamieson T, Silver J, Shuman C, Osmond M, Carroll JC, Jobling R, Laberge AM, Aronson M, Liston E, Lerner-Ellis J, Marshall C, Brudno M, Pham Q, Rudzicz F, Cohn R, Mamdani M, Smith M, Shastri-Estrada S, Seto E, Thorpe K, Ungar W, Hayeems RZ, Bombard Y. Genetics Navigator: protocol for a mixed methods randomized controlled trial evaluating a digital platform to deliver genomic services in Canadian pediatric and adult populations. BMJ Open. 2024 Sep 3;14(9):e090084. doi: 10.1136/bmjopen-2024-090084. PMID 39231549